CLINICAL TRIAL: NCT06772181
Title: Multicenter Pilot Study: Leveraging Digital Health to Promote Evidence-Based Physical Activity to Improve Symptoms Among Patients Undergoing Radiation for Breast Cancer (PRO-ACTIVE)
Brief Title: A Digital Health Intervention to Improve Symptoms and Physical Activity During Breast Radiation
Acronym: PRO-ACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1124991; NCI-2024-10340 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (IM@Home program) (Experimental): A subset of patients in the registry will participate in the IM@Home program consisting of 20+ live, virtual mind-body and fitness classes ranging from yoga and tai chi to dance cardio, guided meditation, and music therapy delivered via Zoom over 30-60 minutes. Patients are instructed to complete at least 3 classes per week for 12 weeks.
  Interventions: Behavioral: IM@Home Program; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Interview
- Registry (FitBit, PRO surveys) (Experimental): Patients receive a FitBit activity tracker and complete patient-reported outcomes (PRO) surveys every 2 weeks (Q2W) to monitor fatigue, comorbid symptoms, and physical activity during and immediately after radiation therapy. Patients with presence of self-reported symptoms or physical inactivity at baseline and/or from any Q2W PRO surveys are then invited to participate and register for IM@Home.
  Interventions: Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Interview

INTERVENTIONS:
Behavioral: IM@Home Program — Participate in the IM@Home program delivered via Zoom
  Arms: Intervention (IM@Home program)
Other: Medical Device Usage and Evaluation — Wear a FitBit activity tracker
Other: Questionnaire Administration — Ancillary studies
Other: Interview — Ancillary studies

SUMMARY:
This clinical trial evaluates a digital health intervention for improving symptoms and physical activity among patients with breast cancer undergoing radiation. Cancer-related fatigue is common and strongly associated with quality of life during and after treatment. Increasing emphasis on early symptom detection and management has prompted initiatives to collect patient-reported fatigue from all patients during treatment. Mind-body interventions including physical activity and yoga are recommendations to treat fatigue and comorbid (coexisting) symptoms. Lower socioeconomic status has not only been associated with higher rates of physical inactivity but also with perceptions that it could negatively impact fatigue and quality of life during treatment. A virtual mind-body program called Integrative Medicine at Home (IM@Home) includes cardio fitness and yoga classes in a bundled intervention that has demonstrated decreased fatigue, depression, insomnia, and symptom distress among patients undergoing breast radiation. The IM@Home program may also increase physical activity among patients with breast cancer undergoing radiation.

DETAILED DESCRIPTION:
OUTLINE:

REGISTRY: Patients receive a FitBit activity tracker and complete patient-reported outcomes (PRO) surveys every 2 weeks (Q2W) to monitor fatigue, comorbid symptoms, and physical activity during and immediately after radiation therapy. Patients with presence of self-reported symptoms or physical inactivity at baseline and/or from any Q2W PRO surveys are then invited to participate and register for IM@Home.

INTERVENTION: Patients participate in the IM@Home program consisting of 20+ live, virtual mind-body and fitness classes ranging from yoga and tai chi to dance cardio, guided meditation, and music therapy delivered via Zoom over 30-60 minutes. Patients are instructed to complete at least 3 classes per week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Ability to understand English, or has a caregiver who understands English.
* Ability to understand and willingness to sign a written informed consent document, virtually or in-person.
* Current breast cancer diagnosis.
* Currently receiving radiation with curative intent (including partial breast, whole breast, or regional nodal radiation).

Exclusion Criteria:

* Patients who are non-English speaking that would prevent their participation in IM@Home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible patients that consent to the screening registry (Feasibility) | Up to 6 months
  Will be considered feasible, as designed, if over 50% of eligible patients consent to the screening registry. Will be determined using descriptive statistics.
Proportion of patients with fatigue or other comorbid symptoms enrolling to the Integrative Medicine at Home (IM@Home) virtual intervention (Acceptability) | Up to 6 months
  Will be considered acceptable if 50% of patients reporting fatigue or other comorbid symptoms agree to enroll to the IM@Home intervention. Will be determined using descriptive statistics.
Proportion of patients enrolling in IM@Home virtual intervention that report favorable implementation outcomes (Appropriateness) | At 12 weeks
  Will be assessed using a validated patient-reported outcomes (PRO) scale with responses as agree or completely agree. Will be determined using descriptive statistics.

SECONDARY OUTCOMES:
Proportion of participants meeting guideline recommendations for physical activity | At baseline, 2, 4, 6, 8, 10, and 12 weeks
  Will be assessed using the Godin Leisure Time Exercise Questionnaire. Will be estimated, along with an exact binomial 95% confidence interval, though no formal statistical testing will be performed.
Relationship between self-reported and monitor-based physical activity | At baseline, 2, 4, 6, 8, 10, and 12 weeks
  Will be evaluated graphically via a scatterplot and Bland-Altman plot. Pearson's correlation coefficient will be estimated for descriptive purposes.
Patient-reported fatigue | At baseline, 2, 4, 6, 8, 10, and 12 weeks
  Will be assessed using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events. Will be plotted graphically for all patients, showing those participating in IM@Home compared to those not assigned to IM@Home.
Sleep quality | At baseline, 4, 8, and 12 weeks
  Will be assessed using the Insomnia Severity Index. Paired T-tests will be assessed for significant within-patient differences in insomnia.
Social isolation | At baseline, 6, and 12 weeks
  Will be assessed using the Cancer Loneliness Scale. Paired T-tests will be assessed for significant within-patient differences in social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Gillespie, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - MultiCare Valley Hospital (Spokane), Spokane Valley, Washington

IPD SHARING:
Plan to Share IPD: No